CLINICAL TRIAL: NCT05228860
Title: Addressing Diabetes by Elevating Access to Nutrition: the ADELANTE Study
Brief Title: Addressing Diabetes by Elevating Access to Nutrition
Acronym: ADELANTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: La Clínica de La Raza Inc. (Other); National Institutes of Health (NIH) (NIH); Dig Deep Farms (Unknown); Yeyi Organics (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lisa Goldman Rosas, Principal Investigator, Assistant Professor, Department of Health Research and Policy (Epidemiology) and Medicine (Primary Care and Population Health) Faculty Director, Office of Community Engagement Stanford School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 62283; 1R01MD016738-01 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Obesity; Lifestyle, Healthy
Keywords: food insecurity; community health worker; health coach; weight loss; HbA1c; T2DM; glycemic control; multilevel
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive household food deliveries and intensive lifestyle intervention OR to a waitlist control group who only receives the household food deliveries (after a 6 month wait). Both groups will be followed for 12 months. Both groups will continue usual primary care for their diabetes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will know which group they have been randomized to. The investigator and statistician will not know to which group a participant belongs. Group identifiers will be removed prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food and Lifestyle Intervention Group (Experimental): The Food and Lifestyle Intervention Group will receive weekly household deliveries of healthy food as well as a lifestyle intervention (called Vida Sana) that will be delivered via Zoom and facilitated by a trained bilingual/bicultural health coach.
  Interventions: Behavioral: Vida Sana (a Group Lifestyle Intervention); Behavioral: Supplemental Healthy Food Deliveries
- Waitlist Control Group (Experimental): The waitlist control will continue usual care with no intervention for 6 months. To balance rigor with ethical considerations, they will receive the healthy food box deliveries after a 6 month waiting period.
  Interventions: Behavioral: Supplemental Healthy Food Deliveries

INTERVENTIONS:
Behavioral: Vida Sana (a Group Lifestyle Intervention) — Vida Sana is a Group Lifestyle intervention that has been shown to be effective among patients with type 2 diabetes (T2DM). Vida Sana includes 23 group sessions with a trained health coach:
  * Months 1-4: 1 family-wide orientation + 12 weekly sessions
  * Months 5-6: 4 bimonthly group sessions
  * Months 7-12: 6 monthly group sessions
  All regular primary care and diabetes care will remain as usual.
  Arms: Food and Lifestyle Intervention Group
Behavioral: Supplemental Healthy Food Deliveries — Participants will receive 12 weeks of weekly food deliveries from Dig Deep Farms.
  Each delivery will include a selection of seasonal fresh vegetables and a rotation of either a whole grain or a whole-grain food (3+ grams of fiber/serving). Whole grains will include brown rice, oatmeal, barley, quinoa; whole grain foods will include cereal, pasta, tortillas, bread, crackers. Delivery sizes will be scaled to the three corresponding household sizes: 2-3 people; 4-5 people; or 6 or more people.
  Food will be delivered by Dig Deep Farms, which already has an established food subscription delivery system.
  (Control group participants will receive the same delivery schedule, but delayed to begin 6 months after their study enrollment.)

SUMMARY:
The goal of ADELANTE is to determine whether a multi-level intervention to improve household food insecurity and glycemic control is effective for Latino patients with diabetes.

Specifically, ADELANTE aims to

1. determine whether weekly household food delivery plus an intensive lifestyle intervention is more effective than usual care for improving glycemic control (HbA1c) at 6 months,
2. examine the effects of the multi-level intervention on = household food insecurity, dietary behaviors, and psychosocial outcomes, and
3. assess the future potential for implementation and dissemination of this multi-level intervention in primary care settings.

DETAILED DESCRIPTION:
Participants and up to two of their household members will be randomized to one of two groups:

1. healthy food box home delivery for 12 weeks plus a 12-month remotely delivered lifestyle behavioral intervention, Vida Sana, which incorporates family members and is aligned with Latino cultural values, or
2. a wait list control group who will receive the food box deliveries 6 months later (but not the Vida Sana intervention).

The first 6 months will evaluate the effects of receiving Vida Sana plus food delivery versus being randomized to control (no intervention); the final 6 months will evaluate receiving food delivery with versus without Vida Sana.

VIDA SANA (intervention arm):

The Vida Sana intervention is a cultural adaptation of Group Lifestyle Balance, a 12-month group program in turn adapted from the NIH/NIDDK-supported Diabetes Prevention Program (DPP). It has been shown to be effective in promoting clinically significant, modest weight loss and significant improvements in moderate-intensity physical activity. Participants receive a total of 23 group sessions over 12 months with a trained health coach who provides personalized feedback based on self-tracking.

The program emphasizes a) moderate caloric reduction by 500-1,000 calories per day through healthy substitutions, b) incremental increases in moderate physical activity such as brisk walking, and c) behavioral strategies to support successful adoption and maintenance of healthy behaviors. These behavioral strategies include realistic goal setting, fostering social support, and stress management. Study health coaches will also add COVID-specific topics to ensure that participants are equipped to change behavior and manage stress during the pandemic.

FOOD BOXES (intervention arm (immediately) and control arm (6 months later)):

Each healthy food box delivery will include a variety of seasonal produce and a rotation of different whole grain foods (3+ grams of fiber/serving) such as cereal, pasta, tortillas, bread, and crackers. Participants will receive familiar foods as well as (intentionally) unfamiliar items to encourage them to try new foods. All items are also available at low-cost grocery stores so participants can continue to purchase them after the end of the study if they wish. The quantity is scaled to three household sizes. It is intended to supplement a family's food supply and provide opportunities for trying new fiber-rich foods recommended by the Vida Sana intervention.

ELIGIBILITY:
Inclusion Criteria:

* For main study (index/intervention) participants:

  * Age at enrollment: 18+ years
  * Self-identified ethnicity: Hispanic, Latino, Chicano, or Spanish
  * Type 2 diabetes indicated in the electronic health record, e.g. as ICD-10 (International Classification of Diseases) diagnosis code or HbA1c value
  * Have indicated food insecurity according to the screening 2-item Hunger Vital Sign questionnaire
  * Have a Body Mass Index (BMI) => 25
  * Receiving care at our partnering community health centers (e.g., Clinica de la Raza)
  * Currently residing in Alameda or Contra Costa County and not expecting to relocate in the next 6-12 months
  * Have access to phone or computer, email, and some internet for access to remote intervention and completion of follow-up measures
* For household members:

  * Age at enrollment: 12+ years
  * Significantly involved in supporting nutrition in the home including food shopping, preparation, social support for healthy nutrition
  * Willing to complete some questionnaires and attend a single group session.
* For all participants:

  * Able and willing to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent
* Unable to speak, read, or understand English and/or Spanish
* Active substance use or psychotic disorders that would impair participation in a group lifestyle intervention or interfere with follow-up assessments
* Lacking mailing address for delivery of food box
* Planning to relocate out of area within the next 12 months
* Index participant only: Pregnant or planning to become pregnant within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
HgbA1c | Baseline through 12 months post-enrollment
  Study staff will gather fingerstick blood samples for HgbA1c.

SECONDARY OUTCOMES:
nonHDL Cholesterol | Baseline through 12 months post-enrollment
  Study staff will gather fingerstick blood samples for lipid measurements, focusing on non- HDL cholesterol (total minus HDL cholesterol) which is a valuable marker of atherogenic dyslipidemia in diabetic individuals that does not require a fasting state.
Blood Pressure | Baseline through 12 months post-enrollment
  Blood pressure will be measured with an automated cuff with digital readout, or using a traditional sphygmomanometer. A study staff member will conduct the reading. Both systolic and diastolic pressure will be measured.
Change in Body Mass Index (BMI) | Baseline through 12 months post-enrollment
  Weight (kg) and height (cm) will be measured and Body Mass Index (BMI) will be calculated in kg/m^2. Height and weight will be gathered using standardized protocols with a portable scale and stadiometer. At baseline, these will be measured in triplicate for accuracy.
Change in waist-height ratio | Baseline through 12 months post-enrollment
  Waist-height ratio (cm) will be calculated and compared over time. Waist circumference (cm) will be measured at iliac crest. Height (cm) will be measured using standardized protocols.
Pandemic-Related Perceived Stress Scale of COVID-19 (PSS-10-C) | Baseline through 12 months post-enrollment
  Participants will answer 10 questions about their stress related to the pandemic. Scale is made up of 10 items, each of which offers five response options: never, almost never, occasionally, almost always and always. Items 1, 2, 3, 6, 9 and 10 are scored directly from 0 to 4 and items 4, 5, 7 and 8, conversely, from 4 to 0.
  Scores range from 0 to 40, higher scores indicating greater stress.
  The PSS-10-C was adapted from the Scale of Perceived Stress (PSS-10) and independently validated during March 2020 in response to government-mandated COVID-19 quarantines in Columbia (see Campo-Arias et al 2020 in the references section)
Type 2 Diabetes Mellitus Related Stress | Baseline through 12 months post-enrollment
  Diabetes-related stress will be measured using the validated 20-item Problem Areas in Diabetes Survey (PAID) questionnaire. Each item is scored from 0 (not a problem) to 4 (serious problem). The sum of all item scores multiplied by 1.25 gives the total PAID score.
  Scores range from 0 to 100, higher scores reflecting greater emotional distress.
Health-related quality of life (adult participants only) | Baseline through 12 months post-enrollment
  Index participants and adult household members will receive the Short Form-8 (SF-8) questionnaire. SF-8 is an 8-item instrument that measures general aspects of health-related quality of life. Each item covers a different domain: overall health, physical functioning, role physical (difficulties with daily work because of physical pain), bodily pain, vitality, social functioning, mental health, and role emotional (absence from daily activities because of emotional problems).
  Items are assessed individual 5- or 6-point Likert scales, a higher score on each question indicates poorer quality of life in that domain.
Health-related quality of life (adolescent household members only) | Baseline through 12 months post-enrollment
  Instead of the SF-8 (see previous outcome), adolescent household members will receive the Kid-Screen-10, a questionnaire is designed for children ages 8-18 to assess subjective health and psychological, mental, and social well-being.
  Scores range from 10 to 50, with higher scores indicating higher health-related quality of life.
Depression | Baseline through 12 months post-enrollment
  Possible depression will be measured using the Patient Health Questionnaire (PHQ-8), which measures 8 criteria from the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders). Each criteria is scored from "0" (not at all) to "3" (nearly every day). Range is 0-24, higher total score indicates more severe depression.
Depression (index participant only) | Baseline through 12 months post-enrollment
  For index participants, depression will be measured using the Patient Health Questionnaire (PHQ-9), which measures 8 criteria from the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) and a ninth question on suicidal thoughts. Each criteria is scored from "0" (not at all) to "3" (nearly every day). Range is 0-27, higher total score indicates more severe depression.
Anxiety | Baseline through 12 months post-enrollment
  Level of anxiety will be measured using the General Anxiety Disorder-7 (GAD-7). This is a 7 item instrument that uses some of the DSM-V (Diagnostic and Statistical Manual of Mental Disorders) criteria for General Anxiety Disorder along with measuring anxiety symptom severity. Scores range from 0 to 21, higher scores indicate more severe anxiety.
Self-reported Loneliness | Baseline through 12 months post-enrollment
  The validated UCLA 3 item Loneliness Scale will be used. The scale is designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as "hardly ever" (1), "some of the time" (2), or "often" (3).
  Scores range from 3 to 9, higher scores indicate greater levels of loneliness.
Dietary Intake Over 24 Hour Period (index participants only) | Baseline through 12 months post-enrollment
  Index participants will complete three 24-hour diet recalls using the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool. The module includes multiple-pass methodology to capture all foods eaten in the previous 24 hours. A researcher will administer the tool to reduce respondent burden. Output for 24-hour diet recall is extensive, but will include our key dietary outcomes for daily (averaged) intakes of: total vegetables, dark green vegetables, beans/legumes, and whole grains.
  Scores:
  Healthy Eating Index (HEI): 0 to 100, higher indicates greater alignment with healthy dietary guidelines Fruit & vegetable: 0-20 servings/day, higher scores preferred Total calorie intake: 1000-6000 kcal/day Total fat: 0-400 g/day
  Interview method adapted from Conway et al 2004 (see references section).
Dietary Intake (household members only) | Baseline through 12 months post-enrollment
  Household members will be given the 10-item Dietary Screener Questionnaire (DSQ-10). The questionnaire will capture consumption of fruit/vegetables, fiber, whole grains, and added sugars. Scores range from 0 to 100, higher scores indicate more frequent consumption of healthy foods.
  They will also be asked additional questions about whole grain foods, which will be scored the same way. These will be based on the dietary screener developed by Thompson and colleagues (see Thompson et al 2017 in references section).
Diet-Related Behaviors: Food Preferences & Consumption | Baseline through 12 months post-enrollment
  We will create a multi-part questionnaire to assess diet-related behaviors:
  1. Self-efficacy to eat fruits/vegetables will be measured using selected items from the National Cancer Institute's Food Attitudes and Behaviors Survey. Scores range from 7 to 35, higher score indicates greater self-efficacy/confidence in ability to consume fresh fruits and veg.
  2. To assess food preferences, participants will be asked Likert-style questions about specific vegetables and whole grains. Higher score indicates stronger "liking".
  3. To assess healthy food consumption, participants will be asked a series of questions about whether they ate specific whole grain foods in the past 7 days. Higher score indicates more frequent consumption.
  4. There will also be three questions specifically about participants use of brown rice (regular and instant). Individual answers will be compared across time points.
Changes in Diet-Related Behaviors | 6 months through 12 months post-enrollment
  Participants will be asked a series of questions designed by the research team to examine changes in their whole grain and vegetable consumption over the past 6 months. Higher score is generally a better outcome as it indicates increase in consumption of these healthy foods.
Change in physical activity | Baseline through 12 months post-enrollment
  Using the 7-day Physical Activity Recall, each participant will complete a semi-structured interview that estimates their time spent doing physical and sleep activities in the past 7 days.
  Scores are:
  * Leisure time moderate and vigorous physical activity, ranging from 0-1500 min/week, higher scores preferred
  * Total energy expenditure, ranging from 06-60 kcal per kg per day, lower scores preferred.
Food Neophobia Scale (FNS) | Baseline through 12 months post-enrollment
  Comprises 10 items to which responses are given on a seven-point Likert scale ranging from "strongly disagree" to "strongly agree."
  Score ranges from 10 to 70, a higher total score indicates greater food neophobia level and lower tendency to try unfamiliar foods.
Control Over Food Choices | Baseline through 12 months post-enrollment
  Participants will be asked a three part-questionnaire about control and food choices in the past 6 months:
  1. Nutrition security is measured with 4 items about food choice availability. Answers are never, rarely, sometimes, often, or always; higher rankings indicates greater nutrition insecurity. Scores range 0-16.
  2. Healthfulness Control is measured with 2 items about sense of control over what they ate or served to their families. Answers are never, rarely, sometimes, often, or always; higher rankings indicates greater control. Scores range 0-8.
  3. Utilization barriers are measured with 2 items about whether participants are able to select healthy foods and make healthy meals. Each item is ranked never true, sometimes true, often true; higher ranking indicates greater utilization barrier. Scores range 0-8.
Nutrition Security Screener | Baseline through 12 months post-enrollment
  The Nutrition Security Screener (NSS) was developed by Tufts University, Kaiser Permanente, and Los Angeles Department of Public Health. The questionnaire contains 14 questions, divided into two sections:
  1. "How hard was it for you or your household to regularly get and eat healthy foods?" Answers are "very hard" (0) , "hard" (1), "somewhat hard"(2) "not very hard" (3) and "not hard at all." (4).
  2. Participants are asked rate 13 different barriers to being able to eat or prepare healthy meals. Each item is ranked "very little or not at all", "somewhat" or "a great deal."
  Question 1 will be scored on a scale of 1-4 to indicate if food security is very low, low, marginal, or secure. Measure designers have not validated a scale for question 2, so it will be analyzed descriptively.
Interest in Community Supported Agriculture (CSA) Programs | Baseline through 12 months post-enrollment
  Community Supported Agriculture (CSA) is a local farm-to-table model where customers can sign up for a subscription with a local farm and receive a weekly box of seasonal fruits and vegetables.
  Participants will be asked a 4 item questionnaire to gauge their experiences with, and interest in, such food boxes, including how much they would be willing to spend for one (e.g. $10-20 per bag). There is no scoring rubric, results are descriptive.
Household Food Insecurity | Baseline through 12 months post-enrollment
  Each participant will complete the USDA's U.S. Household Food Security Survey Module: Six-Item Short Form to measure household food security.
  Raw scores are converted into food security status as follows: 0-1 indicates high or marginal food security, 2-4 indicates low food security, and 5-6 indicates very low food security.
Food Assistance Programs | Baseline through 12 months post-enrollment
  Participants are asked whether their household currently receives (or has received in the past 6 months) various sorts of food assistance, such as:
  * Women, Infants and Children Program (WIC)
  * government food assistance programs known as CalFresh, SNAP (Supplemental Nutrition Assistance Program), EBT (Electronic Benefits Transfer), or food stamps
  * other sources of free food within the last 6 months such as church, food pantry / food bank, soup kitchen, etc, including an open-ended question
  There is no scoring rubric, results are descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goldman Rosas, PhD, MPH, Principal Investigator — Stanford University
Locations (1):
- La Clínica Monument, Concord, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellison B, McFadden B, Rickard BJ, Wilson N. Examining food purchase behavior and food values during the COVID-19 pandemic. Applied Economic Perspectives and Policy. 2021;43(1):58-72. http://dx.doi.org/10.1002/aepp.13118
- [Background] Blair SN, Haskell WL, Ho P, Paffenbarger RS Jr, Vranizan KM, Farquhar JW, Wood PD. Assessment of habitual physical activity by a seven-day recall in a community survey and controlled experiments. Am J Epidemiol. 1985 Nov;122(5):794-804. doi: 10.1093/oxfordjournals.aje.a114163. PMID 3876763
- [Background] Zuazagoitia A, Montoya I, Grandes G, Arietaleanizbeascoa MS, Arce V, Martinez V, Sanchez M, Sanchez A. Reliability and validity of the 7-day Physical Activity Recall interview in a Spanish population. Eur J Sport Sci. 2014;14 Suppl 1:S361-8. doi: 10.1080/17461391.2012.705332. Epub 2012 Jul 25. PMID 24444230
- [Background] Sarkar U, Schillinger D, Lopez A, Sudore R. Validation of self-reported health literacy questions among diverse English and Spanish-speaking populations. J Gen Intern Med. 2011 Mar;26(3):265-71. doi: 10.1007/s11606-010-1552-1. Epub 2010 Nov 6. PMID 21057882
- [Background] Marin G, Gamba RJ. A new measurement of acculturation for Hispanics: The Bidimensional Acculturation Scale for Hispanics (BAS). Hispanic Journal of Behavioral Sciences. 1996;18(3):297-316. http://dx.doi.org/10.1177/07399863960183002
- [Background] Domel SB, Baranowski T, Davis H, Leonard SB, Riley P, Baranowski J. Measuring fruit and vegetable preferences among 4th- and 5th-grade students. Prev Med. 1993 Nov;22(6):866-79. doi: 10.1006/pmed.1993.1078. PMID 8115344
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Conway JM, Ingwersen LA, Moshfegh AJ. Accuracy of dietary recall using the USDA five-step multiple-pass method in men: an observational validation study. J Am Diet Assoc. 2004 Apr;104(4):595-603. doi: 10.1016/j.jada.2004.01.007. PMID 15054345
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Thompson FE, Midthune D, Kahle L, Dodd KW. Development and Evaluation of the National Cancer Institute's Dietary Screener Questionnaire Scoring Algorithms. J Nutr. 2017 Jun;147(6):1226-1233. doi: 10.3945/jn.116.246058. Epub 2017 May 10. PMID 28490673
- [Background] Calloway EE, Carpenter LR, Gargano T, Sharp JL, Yaroch AL. Development of new measures to assess household nutrition security, and choice in dietary characteristics. Appetite. 2022 Dec 1;179:106288. doi: 10.1016/j.appet.2022.106288. Epub 2022 Aug 29. PMID 36049571
- [Background] Campo-Arias A, Pedrozo-Cortes MJ, Pedrozo-Pupo JC. Pandemic-Related Perceived Stress Scale of COVID-19: An exploration of online psychometric performance. Rev Colomb Psiquiatr (Engl Ed). 2020 Oct-Dec;49(4):229-230. doi: 10.1016/j.rcp.2020.05.005. Epub 2020 Jul 17. No abstract available. PMID 33328014
- [Derived] Radtke MD, Chen WT, Xiao L, Rodriguez Espinosa P, Orizaga M, Thomas T, Venditti E, Yaroch AL, Zepada K, Rosas LG, Tester J. Addressing diabetes by elevating access to nutrition (ADELANTE) - A multi-level approach for improving household food insecurity and glycemic control among Latinos with diabetes: A randomized controlled trial. Contemp Clin Trials. 2024 Nov;146:107699. doi: 10.1016/j.cct.2024.107699. Epub 2024 Sep 23. PMID 39322114